CLINICAL TRIAL: NCT03476655
Title: Clinical Outcomes of CLL and MCL Patients Treated With Ibrutinib: An Observational Retrospective Medical Chart Review From India
Brief Title: Clinical Outcomes of Chronic Lymphocytic Leukemia (CCL) and Mantle Cell Lymphoma (MCL) Participants Treated With Ibrutinib: A Medical Chart Review From India
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108441; 54179060LYM4007 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Chronic Lymphocytic Leukemia (CLL): This study will collect retrospective data on effectiveness and outcome parameters for participants of CLL being managed with ibrutinib in the clinical practice. The primary data source for this observational study will be the medical records of each enrolled participant.
  Interventions: Drug: Ibrutinib
- Participants with Mantle Cell Lymphoma (MCL): This study will collect retrospective data on effectiveness and outcome parameters for participants of MCL being managed with ibrutinib in the clinical practice. The primary data source for this observational study will be the medical records of each enrolled participant.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — No study treatment will be administered as a part of this study. Participants in this observational study with confirmed diagnosis of CLL and MCL receiving ibrutinib treatment before 30 April 2018 in routine clinical practice settings will be observed.
  Other Names: IMBRUVICA

SUMMARY:
The purpose of this study is to describe the effectiveness (overall response rate [ORR] and time to progression [TPP]) of Ibrutinib therapy in participants with chronic lymphocytic leukemia (CLL) and mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL) or Mantle Cell Lymphoma (MCL)
* CLL or MCL participants being newly initiated on Imbruvica treatment (ibrutinib capsule 140 mg) based on independent clinical judgment of treating physicians

Exclusion Criteria:

- Any contraindications to ibrutinib use according to the current version of the Prescribing information in India

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population include chronic lymphocytic leukemia (CLL) or mantle-cell lymphoma (MCL) participants treated with ibrutinib per routine clinical care before 30 April 2018 in India and who have progressed on at least one prior line of therapy or CLL participants with deletion 17p (deletions in the short arm of chromosome 17).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 14 months
  ORR is defined as achievement of complete response (CR) or partial response (PR) per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 guidelines for Chronic Lymphocytic Leukemia (CLL) and Mantle-cell Lymphoma (MCL). CR is defined as resolution of enlarged lymph nodes, spleen and liver; normalization of blood counts (neutrophils, hemoglobin, platelets); no residual CLL/MCL detectable in the bone marrow. PR is defined as 50 percent (%) or more reduction in size of enlarged lymph nodes, liver or spleen; 50% or more improvement of blood counts; 50% or more reduction in the blood lymphocyte count.
Time to Progression (TTP) | Up to 14 months
  Time to progression will be reported for the observed participants receiving ibrutinib. TTP is defined as the period from study entry until objective disease progression (time from the date of randomization until disease progression or death due to progression, whichever occur first).
Percentage of Participants with Complete Response (CR) | Up to 14 months
  Percentage of participants with CR will be reported. CR is defined as resolution of enlarged lymph nodes, spleen and liver; normalization of blood counts (neutrophils, hemoglobin, platelets); no residual CLL/MCL detectable in the bone marrow.
Percentage of Participants with Partial Response (PR) | Up to 14 months
  Percentage of participants with PR will be reported. PR is defined as 50 percent (%) or more reduction in size of enlarged lymph nodes, liver or spleen; 50% or more improvement of blood counts; 50% or more reduction in the blood lymphocyte count.
Percentage of Participants with Stable Disease (SD) | Up to 14 months
  Percentage of participants with SD will be reported. Participants who have not achieved a CR or a PR, and who have not exhibited progressive disease will be considered to have stable disease.
Percentage of Participants with Progressive Disease (PD) | Up to 14 months
  Percentage of participants with PD will be reported. PD is defined as 50% or more increase in lymph nodes or the appearance of new enlarged lymph nodes; 50% or more increase in the size of the spleen or liver; 50% or more increase in blood lymphocyte count.

SECONDARY OUTCOMES:
Median time to Response with Ibrutinib | Up to 14 months
  Median time to response with ibrutinib in CLL and MCL participants will be reported. Time to response is defined as the time from start of ibrutinib therapy until objective response (CR or PR assessed by the investigator, based on physical examinations, CT scans, laboratory results, and bone marrow examinations, according to the modified 2008 IWCLL response criteria).
Change from Baseline in Hemoglobin Levels | Baseline up to 14 months
  Change from baseline in blood hemoglobin level will be reported.
Change from Baseline in Platelet Counts | Baseline up to 14 months
  Change from baseline in blood platelet counts will be reported.
Number of Participants with Response to Ibrutinib by Prior Lines of Therapy | Up to 14 months
  Number of participants, who progresses on at least one prior line of therapy, with response to ibrutinib will be reported.
Number of Participants with Hematological and Non-hematological Adverse Drug Reactions (ADR) | Up to 14 months
  Number of participants with hematological and non-hematological ADR will be reported. An adverse drug reaction (ADR) is defined as a response to a medicinal (investigational or non-investigational) product that is noxious and unintended. The phrase "response to a medicinal product" means that a causal relationship between a medicinal product and an adverse event is possible, probable or very likely.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (8):
- India (8):
  - Apollo Hospitals International Limited, Ahmedabad
  - Healthcare Global (HCG) Hospital, Bangalore
  - Fortis Memorial Research Institute, Gūrgaon
  - Basavatarakam Indo-American Hospital, Hyderabad
  - Bhagwan Mahaveer Hospital & Research Centre, Jaipur
  - Tata Medical Center, Kolkata
  - All India Institute of Medical Sciences, New Delhi
  - Yashoda Hematology Clinic, Pune